CLINICAL TRIAL: NCT02099435
Title: A Prospective Observational Cohort Study of Hemospray for Lower Gastrointestinal Hemorrhage (APPROACH LGI)
Brief Title: Study of Hemospray for Lower Gastrointestinal Hemorrhage
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-007
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Colonic Diverticula; Angiodysplasia; Colonic Polyp
Keywords: Gastriointestinal; Lower gastriointestinal; Digestive; Hemostasis; Recurrent bleeding; Hemospray
MeSH Terms: conditions — Diverticulum, Colon; Angiodysplasia; Colonic Polyps; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemospray to treat lower GI bleeds
  Interventions: Device: Hemospray

INTERVENTIONS:
Device: Hemospray — The Hemospray™ device comes in a 7F kit and a 10F kit. Each kit includes two 220 cm Teflon application catheters, a handle with CO2 cartridge and a syringe containing approximately 20 g of the Hemospray™ material. Hemospray™ is a proprietary inorganic mineral powder that acts as a mechanical barrier when sprayed over a bleeding lesion and the surrounding mucosa.

SUMMARY:
This study is to evaluate the performance of Hemospray for the teatment of nonvariceal lower gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patient in which Hemospray is used to treat an endoscopically confirmed nonvariceal lower GI bleed requiring hemostasis

Exclusion Criteria:

* Less than 19 years old
* Unwilling or unable to sign and date the informed consent
* Pregnant, lactating or planning to become pregnant within 30 days of the procedure
* Contraindicated to undergo colonoscopy

Medical/Endoscopic Exclusion Criteria

* Actual or suspected lower GI perforation or fistula
* Bleeding originating from inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
* Actual or suspected ischemic colitis or infectious colitis
* Unable to visualize site of active bleeding (such as suspected diverticular bleed where source is unable to be identified)
* Unable to treat active site of bleeding (e.g., bleeding site cannot be reached by the colonoscope)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11-06 (Actual); Study Completion 2016-11-06 (Actual)

PRIMARY OUTCOMES:
Percentage of device related adverse events | 30 days

SECONDARY OUTCOMES:
Percentage of recurrent bleeding that occurs outside the blood vessel | 30 days
Percentage of hemostasis of lower GI bleeds originating from multiple sources | 30 days
All cause mortality | 30 days
  Mortality within 30 days of index procedure

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Hotel Dieu Hospital, Kingston, Ontario
  - Montreal General Hospital - McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Hookey L, Barkun A, Sultanian R, Bailey R. Successful hemostasis of active lower GI bleeding using a hemostatic powder as monotherapy, combination therapy, or rescue therapy. Gastrointest Endosc. 2019 Apr;89(4):865-871. doi: 10.1016/j.gie.2018.10.029. Epub 2018 Oct 26. PMID 30612959